CLINICAL TRIAL: NCT04393805
Title: Heparins for Thromboprophylaxis in COVID-19 Patients: HETHICO Study in Veneto
Acronym: HETHICO
Status: Completed | Type: Observational
Sponsor: Quovadis Associazione (Other)
Collaborators: University of Padova (Other)
Responsible Party: Sponsor
Other Study IDs: HETHICO
Record Dates: First submitted 2020-05-16; First posted 2020-05-19 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: COVID-19; Hypercoagulability
Keywords: COVID-19 pandemic; Hypercoagulability state; Thromboprophylaxis; Heparin
MeSH Terms: conditions — COVID-19; Thrombophilia | interventions — Heparin, Low-Molecular-Weight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes

GROUPS / COHORTS (2):
- MED-Cohort: Patients hospitalized for SARS-COVID-2 infection in a medical ward
  Interventions: Drug: Low Molecular Weight Heparin
- ICU-Cohort: Patients hospitalized for SARS-COVID-2 infection in a sub-intensive or intensive care unit
  Interventions: Drug: Low Molecular Weight Heparin

INTERVENTIONS:
Drug: Low Molecular Weight Heparin — Thromboprophylaxis with Low Molecular Weight Heparin, mostly enoxaparin
  Other Names: LMWH

SUMMARY:
The HETHICO study aims to collect retrospectively documented clinical information on patients hospitalized in Veneto Region (Italy) for SARS-COVID-2 infection in 2 types of settings, medical environment (COORTE MED), and intensive / sub-intensive (COORTE ICU), to assess the safety and possible efficacy of the anticoagulant treatments used for thromboprophylaxis, or in preventing thrombotic complications related to hospitalization from COVID-19.

DETAILED DESCRIPTION:
The HETHICO study aims to collect retrospectively documented clinical information on patients hospitalized in Veneto Region (Italy) for SARS-COVID-2 infection in 2 types of settings, medical environment (COORTE MED), and intensive / sub-intensive (COORTE ICU), to assess the safety and possible efficacy of the anticoagulant treatments used for thromboprophylaxis, or in preventing thrombotic complications related to hospitalization from COVID-19.

Furthermore, the possible association between the observed clinical evolution and the type of antithrombotic prophylaxis performed (class of drug and dose intensity) will be assessed in a large cohort of patients hospitalized in the various participating hospitals in the Veneto region and observed with follow-up. in the short term, gathering information on:

Clinical outcomes, Survival, Concomitant pathologies, Adverse events of anticoagulant drugs, Interactions with other concomitant drugs, and Risk factors.

The collected data, suitably anonymized, will be used to produce scientific works, the standardization of care paths, and the planning of targeted training events.

ELIGIBILITY:
Inclusion Criteria:

* proved SARS-COVID-2 infection

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects of both sexes, aged 18 years or older (no maximum age of inclusion) will be eligible for this study, who have been hospitalized in the participating Operating Units (Centers) of Veneto Region Hospitals with infection SARS-COVID-2.
Sampling Method: Non-Probability Sample
Enrollment: 744 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-02-26 (Actual); Study Completion 2021-02-26 (Actual)

PRIMARY OUTCOMES:
Bleeding | 28 days
  Collect and evaluate in real-life the safety data of the anti-coagulant treatments used by estimating the incidence of bleeding complications during hospitalization.
Thrombosis | 28 days
  Collect and evaluate in real-life the efficacy data of the anti-coagulant treatments used by estimating the incidence of deep vein thrombosis and/or pulmonary embolism during hospitalization.
Mortality | 28 days
  Collect and evaluate in real-life the data by estimating incidence of intra-hospital death.

SECONDARY OUTCOMES:
Worsening | 28 days
  clinical worsening with transfer to the intensive/sub-intensive ward
LOS | 60 days
  length of stay

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Simioni, Prof., Principal Investigator — Department of Medicine, University of Padua (I)
Locations (1):
- Giuseppe Camporese, Padua, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Flumignan RL, Civile VT, Tinoco JDS, Pascoal PI, Areias LL, Matar CF, Tendal B, Trevisani VF, Atallah AN, Nakano LC. Anticoagulants for people hospitalised with COVID-19. Cochrane Database Syst Rev. 2022 Mar 4;3(3):CD013739. doi: 10.1002/14651858.CD013739.pub2. PMID 35244208
- [Derived] Flumignan RL, Tinoco JDS, Pascoal PI, Areias LL, Cossi MS, Fernandes MI, Costa IK, Souza L, Matar CF, Tendal B, Trevisani VF, Atallah AN, Nakano LC. Prophylactic anticoagulants for people hospitalised with COVID-19. Cochrane Database Syst Rev. 2020 Oct 2;10(10):CD013739. doi: 10.1002/14651858.CD013739. PMID 33502773